CLINICAL TRIAL: NCT03385577
Title: Feasibility, Acceptability, and Efficacy of a Yoga Intervention for Distress in Women With Gynecologic, Gastrointestinal, or Thoracic Cancer
Brief Title: Yoga for Psychological Distress in Gynecologic, Gastrointestinal, or Thoracic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB201700079; OCR16587 (Other: OnCore)
Record Dates: First submitted 2017-12-20; First posted 2017-12-28 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Gynecologic Cancer; Adjustment; Gastrointestinal Cancer; Thoracic Cancer
Keywords: Gastrointestinal (GI); Fear of Cancer Recurrence (FCR)
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Yoga Intervention (Experimental): The intervention, "Stilling the Waters of Uncertainty: A yoga program for women with gynecologic, gastrointestinal (GI), or thoracic cancer," is a 10-week, manualized, group yoga program. Sessions are 60 minutes in duration, once a week, across the course of 10 weeks. The 10-week program is comprised of five modules, each of which will take two sessions to complete: (1) Getting Started, (2) Cultivating a Mindful Attitude, (3) Self-Care and Compassion, (4) Finding Peace and Acceptance, and (5) The Power of the Present Moment.
  Interventions: Behavioral: Stilling the Waters of Uncertainty: A yoga program for women with gynecologic, gastrointestinal (GI), or thoracic cancer

INTERVENTIONS:
Behavioral: Stilling the Waters of Uncertainty: A yoga program for women with gynecologic, gastrointestinal (GI), or thoracic cancer — 'Stilling the waters,' the prominent theme of this program, is drawn from the core principle in yogic philosophy. It uses breath techniques and physical postures to cultivate inner peace and an ability to live in the present moment. The emphasis on stilling the fluctuations of uncertainty is a direct allusion to the intrusive and inherently unknown future, which characterizes the core experience of Fear of Cancer Recurrence (FCR). This is especially true among gynecologic, gastrointestinal (GI), or thoracic cancer patients for whom the likelihood of recurrence is quite high. An additional motif throughout the program is the lotus flower. The symbolic importance of the lotus in yogic culture is due to its requiring thick muddy waters for ideal growth. The metaphor of cancer as the muddy waters will be used to cultivate benefit-finding and acceptance regarding the mental and physical challenges participants endured during their initial diagnosis and treatment.

SUMMARY:
This study will test the feasibility and acceptability of a yoga program for women with gynecologic, gastrointestinal (GI), or thoracic malignancies. This study will pilot an integrative yoga intervention that combines Western psychotherapeutic approaches with classic yogic philosophy to reduce emotional distress among women undergoing treatment for gynecologic, gastrointestinal (GI), or thoracic cancer and provide a comprehensive approach to stress management across the cancer care continuum.

DETAILED DESCRIPTION:
Gynecologic cancers are malignancies of the female reproductive tract that affect over 70,000 women per year. Treatments for gynecologic cancer often result in numerous physical and emotional side effects that affect long-term adjustment, such as anxiety, depression, low self-esteem, sexual dysfunction, difficulties with fertility, and surgically-induced menopause. Even when initial treatments are successful, gynecologic cancers have a high recurrence rate that can reach nearly 80% among those with ovarian cancer. Fear of Cancer Recurrence (FCR) is described as one of the largest unmet psychological needs among gynecologic cancer patients and is associated with psychological distress, increased health care utilization, and functional impairment. Few studies have examined interventions designed to manage symptoms of FCR, which leaves a significant gap in the literature regarding treatment of this prominent psychosocial problem. Cancer patients report growing use of integrative medicine therapies (e.g., yoga, acupuncture, massage) to manage unmet physical and emotional needs related to their disease and treatment. The current study will take advantage of this trend in supportive oncology to investigate the feasibility and acceptability of a novel intervention program created specially to address FCR among women with gynecologic cancer. Patients will be recruited from the UF Health/Shands Hospital Gynecology Oncology Clinic and Medical Oncology clinic and invited to participate in a 10-week, manualized, small group yoga course. Psychoeducation modules, meditation training, and gentle yoga poses will be integrated into a comprehensive program focused on managing the psychosocial concerns of newly diagnosed gynecologic cancer patients. Findings from this research will contribute to the existing literature on FCR and knowledge regarding the use of integrative medicine techniques for addressing unmet psychological needs among gynecologic cancer patients. If the intervention is deemed feasible and acceptable, future research may explore ways in which this manualized yoga program compares to other psychosocial treatments for managing FCR and other forms of emotional distress in women with cancer.

ELIGIBILITY:
Inclusion Criteria:

* Presence of newly diagnosed
* pathology-confirmed
* (a) gynecologic cancer (e.g., cancer of the ovaries, cervix, endometrium, fallopian tubes), any stage, or
* (b) borderline ovarian tumor, Stage II-III
* Undergoing (or have recently undergone) surgery and/or active cancer treatment (e.g., chemotherapy, radiation, a combination of these treatments and/or another form of cancer treatment)
* Able to read and write in English

Exclusion Criteria:

* History of gynecologic cancer or other cancer diagnosis (excluding basal cell or squamous cell carcinomas of the skin)
* Current, severe, uncontrolled psychopathology (e.g., symptomatic Bipolar Disorder with a manic or depressive episode in the last six months, psychotic symptoms or disorder, or documented personality disorder)
* History of dementia or other neurocognitive disorder that may interfere with participants' ability to adhere to study procedures
* Poor performance status as determined by a Karnofsky Status Score < 60,
* For those with any childbearing potential (i.e., 18 - 62 years of age, have intact reproductive organs, and/or have not yet started chemotherapy or radiation therapy): self-reported current pregnancy, possible pregnancy, or efforts to become pregnant
* History of regular or immersive yoga practice in the last five years defined as attending at least once weekly yoga classes for at least 6 consecutive months at any point in the prior 5 years

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2022-11-14 (Actual)

PRIMARY OUTCOMES:
Feasibility of the proposed yoga program - Study enrollment rate | Pre-Intervention (Baseline) to Post-Intervention (Ten Weeks After Baseline)
  Patients will complete the majority (80%) of study activities as measured by five empirically-driven indicators of feasibility.
Feasibility of the proposed yoga program - Intervention session attendance | Pre-Intervention (Baseline) to Post-Intervention (Ten Weeks After Baseline)
  Patients will complete the majority (80%) of study activities as measured by five empirically-driven indicators of feasibility.
Feasibility of the proposed yoga program - Adherence to homework assignments | Pre-Intervention (Baseline) to Post-Intervention (Ten Weeks After Baseline)
  Patients will complete the majority (80%) of study activities as measured by five empirically-driven indicators of feasibility.
Feasibility of the proposed yoga program - Retention through follow-up assessment (i.e., individuals who complete all components of the study) | Pre-Intervention (Baseline) to Post-Intervention (Ten Weeks After Baseline)
  Patients will complete the majority (80%) of study activities as measured by five empirically-driven indicators of feasibility.
Feasibility of the proposed yoga program - Safety (i.e., adverse events) | Pre-Intervention (Baseline) to Post-Intervention (Ten Weeks After Baseline)
  Patients will complete the majority (80%) of study activities as measured by five empirically-driven indicators of feasibility
Program Acceptability- Relevance of the intervention to their lives | Pre-Intervention (Baseline) to Post-Intervention (Ten Weeks After Baseline)
  The majority of patients (80%) will rate five key dimensions of the intervention on a Likert scale as "Very" or "Extremely" acceptable.
Program Acceptability- the Utility of the intervention to participants | Pre-Intervention (Baseline) to Post-Intervention (Ten Weeks After Baseline)
  The majority of patients (80%) will rate five key dimensions of the intervention on a Likert scale as "Very" or "Extremely" acceptable.
Program Acceptability- Satisfaction/Enjoyment of the intervention | Pre-Intervention (Baseline) to Post-Intervention (Ten Weeks After Baseline)
  The majority of patients (80%) will rate five key dimensions of the intervention on a Likert scale as "Very" or "Extremely" acceptable.
Program Acceptability - Clarity/Ease of the intervention for participants | Pre-Intervention (Baseline) to Post-Intervention (Ten Weeks After Baseline)
  The majority of patients (80%) will rate five key dimensions of the intervention on a Likert scale as "Very" or "Extremely" acceptable.
Program Acceptability - Plan to continue intervention exercises after completion of the study | Pre-Intervention (Baseline) to Post-Intervention (Ten Weeks After Baseline)
  The majority of patients (80%) will rate five key dimensions of the intervention on a Likert scale as "Very" or "Extremely" acceptable.

SECONDARY OUTCOMES:
Fear of Cancer Recurrence (FCR) | Pre-Intervention (Baseline) to Post-Intervention (Ten Weeks After Baseline)
  This measure will access participants' Fear of Cancer Recurrence (FCR), which includes cognitive, behavioral, and emotional experiences related to worries that their cancer will return.
Cancer-Related Distress | Pre-Intervention (Baseline) to Post-Intervention (Ten Weeks After Baseline)
  The Distress Thermometer will be used to assess cancer-related distress. This measure is designed to assess self-efficacy regarding distress and symptom management while facing a cancer diagnosis. Domains assessed include maintenance of activity and independence, seeking and understanding medical information, stress management, coping with treatment side effects, maintaining a positive attitude, engaging in emotion regulation, and seeking support.
State and Trait Anxiety | Pre-Intervention (Baseline) to Post-Intervention (Ten Weeks After Baseline)
  Anxiety will be assessed with the State Trait Anxiety Inventory (STAI) Assesses state /trait anxiety symptoms on 4 pt. likert scale. Medium: May indicate anxiety disorder
Depressive Symptoms | Pre-Intervention (Baseline) to Post-Intervention (Ten Weeks After Baseline)
  Depressive symptoms will be assessed with the Beck Depression Inventory - Second Edition (BDI-2) - high score Suicidal Behavior

CONTACTS AND LOCATIONS:
Overall Officials: Deidre B. Pereira, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hanvey GA, Padron A, Kacel EL, Cartagena G, Bacharz KC, McCrae CS, Robinson ME, Waxenberg LB, Antoni MH, Berry RB, Schultz GS, Castagno J, Pereira DB. Accrual and retention of diverse patients in psychosocial cancer clinical trials. J Clin Transl Sci. 2022 Apr 1;6(1):e45. doi: 10.1017/cts.2022.380. eCollection 2022. PMID 35651964
- [Derived] Hanvey GA, Kacel EL, Bacharz KC, Wilborn AP, Mesa S, McCracken H, Estores IM, Markham MJ, Kaye FJ, Jones D Jr, George TJ, Pereira DB. Proof-of-Concept of an Integrated Yoga and Psychological Intervention in Mitigating Distress Among Diverse Women With Gynecologic, Gastrointestinal, and Thoracic Cancers. Integr Cancer Ther. 2024 Jan-Dec;23:15347354241283113. doi: 10.1177/15347354241283113. PMID 39423043